CLINICAL TRIAL: NCT06103682
Title: LOcally ABLatIve ThErapy for OligopRogressive Lung And Thoracic MalignanciEs (OBLITERATE)
Acronym: OBLITERATE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Megan Daly, MD, Principal Investigator, University of California, Davis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCDCC313
Record Dates: First submitted 2023-10-19; First posted 2023-10-27 (Actual); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Non-small Cell Lung Cancer; Oligoprogressive; Small-cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Ablative local therapy (Experimental): Stereotactic ablative radiotherapy (SABR) or interventional radiology (IR) ablation therapy
  Interventions: Device: Ablative local therapy

INTERVENTIONS:
Device: Ablative local therapy — Stereotactic ablative radiotherapy (SABR) or interventional radiology (IR) ablation therapy

SUMMARY:
This is a phase 2 pragmatic study that evaluates the clinical benefit of continuing systemic therapy with the addition of locally ablative therapies for oligo-progressive solid tumors as the primary objective. The primary outcome measure is the time to treatment failure (defined as time to change in systemic failure or permanent discontinuation of therapy) following locally ablative therapy.

DETAILED DESCRIPTION:
This is a phase 2 pragmatic study at a single site that evaluates the clinical benefit of continuing systemic therapy with the addition of locally ablative therapies for oligo-progressive solid tumors as the primary objective. The primary endpoint is disease control at 3 months, defined as continuation in systemic cancer therapy without any changes or permanent discontinuation for 3 months following first day of ablative local therapy. Participants will receive ablative local therapy per standard practices in addition to their systemic therapy and will be followed for up to 5 years following ablative local therapy. Participants will be assigned stereotactic ablative radiotherapy (SABR) or interventional radiology (IR) ablation therapy per the discretion of treating radiation oncologist and/or interventional radiologist.

ELIGIBILITY:
Inclusion Criteria:

1. Must have one of the following histologically and/or biochemically confirmed genitourinary malignancies:

   1. Cohort A: Non-small cell cancer
   2. Cohort B: Small cell cancer
2. Provision of signed and dated informed consent form.
3. Stated willingness to comply with all study procedures and availability for the duration of the study.
4. Age ≥18 years at time of consent.
5. Currently on systemic therapy and a candidate to continue their current line of systemic therapy with no more than a planned 30-day break to allow for local ablative therapy.
6. ≥ 1 line of systemic therapy for metastatic disease with ≥ 3 months of clinical benefit on most recent line of systemic therapy prior to the development of new metastatic lesions. [Clinical benefit: Treating provider assessment that majority of the tumor burden is stable on current systemic treatment and not requiring an immediate change in systemic treatment]
7. ≤ 5 progressing or new metastatic lesions.
8. All progressing or new metastatic lesions can be safely treated with locally ablative therapies at discretion of treating radiation oncologist and/ interventional radiologist.

Exclusion Criteria:

1. Medical comorbidities precluding locally ablative therapies.
2. History of treatment related toxicities that limit or prohibit application of locally ablative therapies.
3. Progressing intracranial lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-10-05 (Actual); Primary Completion 2025-12-05 (Estimated); Study Completion 2031-01-05 (Estimated)

PRIMARY OUTCOMES:
Number of participants with controlled disease | 3 months from the first day of ablative local therapy
  Number of participants with controlled disease at 3 months, defined as continuation in systemic cancer therapy without any changes or permanent discontinuation for 3 months following first day of ablative local therapy

SECONDARY OUTCOMES:
Number of participants experiencing grade ≥ 3 adverse events attributable to ablative local therapy | Up to 2 years from the first day of ablative local therapy
  Number of participants experiencing grade ≥ 3 adverse events (except for hematologic and electrolyte abnormalities) attributable to ablative local therapy occurring up to 2 years from the first day of ablative local therapy
Median overall survival | Up to 1 year from the first day of ablative local therapy
  Median overall survival stratified by primary tumor type
Time to treatment failure | Up to 1 year from the first day of ablative local therapy
  Time to treatment failure, defined as time to change in systemic therapy or permanent discontinuation of cancer therapy

CONTACTS AND LOCATIONS:
Overall Officials: Megan Daly, MD, Principal Investigator — University of California, Davis
Locations (1):
- University of California, Davis, Sacramento, California, United States